CLINICAL TRIAL: NCT04478058
Title: Feasibility and Effectiveness of Delivering Cognitive Behaviour Therapy Through Online Psychotherapy Tool (OPTT) for Depression
Brief Title: Feasibility and Effectiveness of Delivering CBT Through OPTT for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Nazanin Alavi (Other)
Collaborators: Online PsychoTherapy Clinic (Other)
Responsible Party: Sponsor-Investigator, Dr. Nazanin Alavi, Principal Investigator, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSIY-563-17
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression; e-CBT; Online Psychotherapy; Cognitive Behavioural Therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Participants will be offered to take part in either live or online Cognitive Behavioural Therapy for a 12 week period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-CBT (Experimental): Weekly e-CBT sessions will occur through Online Psychotherapy Tool (OPTT) and consist of slides and interactive therapist videos. Content and format mirrors live CBT. Slides will highlight a different topic each week and include general information, overview of skills, and homework. Homework will be submitted through OPTT and reviewed by administrators with personalized feedback within three days. Weekly homework submission will be mandatory before beginning the next session. DASS 21 and Q-LES-Q-SF questionnaires will be completed at the beginning and end of treatment. After each cycle of e-CBT, patients and healthcare providers involved in e-CBT will be recruited for focus groups once they have completed their 12-week program. Qualitative data will be gathered through 10 focus groups. The focus group prompts will pertain to experience and expectations of service. Patients will be contacted six months after treatment to complete DASS 21 and Q-LES-Q-SF questionnaires.
  Interventions: Behavioral: e-CBT
- Live CBT (Active Comparator): The content and format of live CBT will be mirrored by the e-CBT group over the course of 12 weeks. The sessions will highlight a different topic each week and include general information, an overview of skills, and homework on that topic. Live CBT homework will be reviewed by the CBT group organizer and provided at the beginning of the next CBT session. Weekly homework submission for feedback will be mandatory before being eligible for the next session. DASS 21 and Q-LES-Q-SF questionnaires will be completed at the beginning and end of treatment for both live and e-CBT. All live and e-CBT patients will be contacted six months after the completion of their CBT to complete final DASS 21 and Q-LES-Q-SF questionnaires. This will allow for the examination of the longevity of e-CBT compared to live CBT.
  Interventions: Behavioral: Live CBT

INTERVENTIONS:
Behavioral: Live CBT — Weekly in-person Cognitive Behavioural Therapy
  Arms: Live CBT
Behavioral: e-CBT — Weekly online Cognitive Behavioural Therapy
  Arms: e-CBT

SUMMARY:
Major Depressive Disorder (MDD) is a prevalent and debilitating mental health disorder. Among different therapeutic approaches (e.g., medication, psychotherapy), psychotherapy in the form of cognitive behavioural therapy (CBT) is considered the gold standard treatment for MDD. However, while efficacious, CBT is not readily accessible to many patients in need due to hurdles like stigma, long wait times, high cost, the large time commitment for health care providers, and cultural/geographic barriers. Online delivery of CBT (e-CBT) can effectively address many of these accessibility barriers. Objective: This study aims to investigate the efficacy and feasibility of implementing a digital online psychotherapy clinic for the treatment of MDD. This non-randomized control trial intervention will provide e-CBT for MDD through the Online Psychotherapy Tool (OPTT), a secure, cloud-based, digital mental health platform. Participants (age 18-65 years) will be offered an e-CBT program tailored to MDD over 12 weeks to address their depressive symptoms. Participants will complete pre-designed modules and homework assignments while receiving personalized feedback and asynchronous interaction with a therapist through the platform. Using clinically validated symptomology questionnaires, the efficacy of the e-CBT program will be compared to a group receiving in-person CBT. Questionnaires will be completed at baseline, week 6, week 12, and at a 6-month follow-up. Inclusion criteria include diagnosis of MDD, competence to consent to participate, ability to speak and read English, and consistent and reliable access to the internet. Exclusion criteria include active psychosis, acute mania, severe alcohol or substance use disorder, and/or active suicidal or homicidal ideation. The results from this study can provide valuable information used to develop more accessible and scalable mental health interventions with increased care capacity for MDD, without sacrificing the quality of care.

DETAILED DESCRIPTION:
Study Design For this study, a non-randomized, controlled trial study design will be employed. Qualitative focus groups will be conducted to gather personal demographic information as well as information regarding the feasibility of implementing an online psychotherapy clinic. Additionally, quantitative analyses of e-CBT treatment efficacy will be conducted using standardized and clinically validated symptomology questionnaires. All study procedures have been approved by the Queen's University Health Sciences and Affiliated Teaching Hospitals Research Ethics Board.

Participants Patients (n = 110; 55 e-CBT participants, 55 in-person CBT participants) aged 18-65 years will be recruited at Queen's University from outpatient psychiatry clinic at both Kingston Health Sciences Centre sites (Hotel Dieu Hospital and Kingston General Hospital) as well as Providence Care hospital, family doctors, physicians, clinicians, and self-referrals in Kingston, Ontario, Canada. Once informed consent is provided, participants will be evaluated by a psychiatrist on the research team through secure video appointment to make or confirm a diagnosis of Major Depressive Disorder (MDD) using the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5).

The inclusion criteria for the study include the following: at least 18 years of age at the start of the study, diagnosed with major depressive disorder according to DSM-5 by an attending psychiatrist on the research team, competence to consent to participate, ability to speak and read English, and consistent and reliable access to the internet. Exclusion criteria include active psychosis, acute mania, severe alcohol or substance use disorder, and/or active suicidal or homicidal ideation. If a participant is receiving another form of psychotherapy, they will also be excluded from the study, to avoid any confounding effect on the efficacy of this e-CBT program. If eligible for the study, participants will choose between the e-CBT program (n = 55) or the in-person CBT offered individually through this program at Hotel Dieu Hospital (n = 55).

During the informed consent process, it is explained to all participants that this program is not a crisis resource and that they will not have access to their therapist at all times. In the case of an emergency, participants are directed to the proper resources (e.g., emergency department, crisis lines, etc.) and this event will be reported to the principal investigator of the study.

Procedures The e-CBT care plan consists of 12 weekly sessions of approximately 30 slides and interactive content, delivered through OPTT. The e-CBT module content mirrors in-person group CBT content, including different weekly topics, general information, skill overviews, and homework. The efficacy of the therapeutic content has previously been tested through email administration and shown to significantly reduce depressive symptoms Participants are instructed to go through the content and complete homework at the end of the session which helps them practice skills they learned through that session. Homework is submitted through OPTT and reviewed by the therapist assigned to the participant, who will provide personalized feedback within three days of submission. Therapists have access to pre-designed session-specific feedback templates to use as a basic structure to write their feedback. By doing so, the time needed to respond to each patient is reduced and therefore the number of patients each therapist can handle increases. At the same time, by using a structured format in responding to patients, more standardized quality of care can be assured. The general structure of the feedback template is as follows: -validating the participant's time and effort, -reviewing the event they have used in their homework, -summarizing the previous module's content, and -discussing the participant's homework submission and how they could improve it. In addition to these points, the feedback will have an emphasis on specific content from the participant's submission, reassuring them that their therapist is reading and understanding their challenges. All feedback submissions are finished with a personalized signature from the therapist, helping to develop a rapport between the therapist and the participant. On average, developing this feedback takes a therapist 15-20 minutes per patient. In addition to the weekly feedback, participants have the option to message their therapist through the platform throughout the week regarding any questions or concerns they may have. All technical issues are handled directly through OPTT's technical support team.

Participants in the in-person CBT group will attend weekly sessions at Hotel Dieu Hospital (12 weeks) where they will receive standardized individual (one-on-one) CBT for MDD from a trained therapist. All content covered and skills taught will mirror the e-CBT program. Similar to the e-CBT group, participants will be assigned weekly homework assignments that they will complete during the week and hand-in at the start of their next session. At this time, participants will receive personalized feedback for their previous week's homework from their therapist.

At the end of the study, a few participants and healthcare providers (i.e., 8 participants, 2 providers) are recruited for focus groups. The focus group prompts will pertain to experience and expectations of service during the study and how they think the service could be improved.

Online Module Content Both e-CBT modules and in-person CBT sessions are designed to instill constructive and balanced coping strategies in participants. During the program, we focus on essential thinking and behavioural skills to help the patients become more engaged in day-to-day activities. The focus of the sessions is placed on the connection between thoughts, behaviours, emotions, physical reactions, and the environment. We work on evaluating negative beliefs and thought processes and their relationship with depression. Our goal is to adjust the negative thinking so that participants can think about and adapt to the things that are happening to them. This allows them to adjust the way they behave and think about their problems in a way that is not as negative and replaces those thoughts and behaviours with potentially more realistic and productive ones.

Training All therapists are research assistants hired by the principal investigator. They all undergo training in psychotherapy and additional training from a psychiatrist on the research team before any interaction with participants. During this training, therapists complete feedback on practice homework, which is reviewed by a psychiatrist on the research team to ensure adequate quality of work. All therapists are supervised by the lead psychiatrist, who is an expert in the area of electronically delivered psychotherapy. Feedback is always reviewed by the lead psychiatrist, before submission to the participants.

ELIGIBILITY:
Inclusion Criteria:

* At least 16 years old at the start of the study
* Diagnosed with major depressive disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) by a clinician
* Competence to consent to participate
* Ability to speak and read English
* Consistent and reliable access to the internet

Exclusion Criteria:

* High current suicide risk (score of over 17 points on section C, Suicidality, of MINI)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in symptoms - Patient Health Questionnaire - 9 Item | Week 1, Week 6, Week 12, 6-Month Follow-Up
  Clinical standardized symptom questionnaire. Scale of 0-3, 3 being the worst.
Change in symptoms (Quick Inventory of Depressive Symptomatology) | Week 1, Week 6, Week 12, 6-Month Follow-Up
  Clinical standardized symptom questionnaire. Scale of 0-3, 3 being the worst.
Change in quality of life (Quality of Life Enjoyment and Satisfaction Questionnaire) | Week 1, Week 6, Week 12, 6-Month Follow-Up
  Clinical standardized symptom questionnaire. Scale of 1-5, 1 being the worst.

SECONDARY OUTCOMES:
Qualitative Analysis - Healthcare Provider Experience | Week 12 (Post-Treatment)
  Focus groups for healthcare providers who will be asked about feasibility of providing the e-psychotherapy program, how it compares to in-person psychotherapy.
Qualitative Analysis - Participant Experience | Week 12 (Post-Treatment)
  Interviews with participants regarding personal, social, and cultural factors (gender, sexuality, background, supportive resources, structural/social barriers, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin Alavi, MD FRCPC, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Information from this study is confidential and patients' anonymity will be protected. e-CBT participants will have a password-protected encrypted file through the OPTT. Questionnaires and homework submitted via OPTT can only be accessed by psychiatrists involved in the study and clinicians involved in their care. Data from this research will be saved without mention of any patient names with all patients being identified with a unique identification number in all data from this study. A master file of participant ID numbers and participant names will be maintained in a password-protected encrypted file and destroyed once the study has been completed. Hard copies of patient study files will be stored in locked cabinets and offices and will be available only to clinicians providing treatment and Research Coordinator. Participants will not be identified in any publication or reports.

REFERENCES:
- [Derived] Alavi N, Moghimi E, Stephenson C, Gutierrez G, Jagayat J, Kumar A, Shao Y, Miller S, Yee CS, Stefatos A, Gholamzadehmir M, Abbaspour Z, Shirazi A, Gizzarelli T, Khan F, Patel C, Patel A, Yang M, Omrani M. Comparison of online and in-person cognitive behavioral therapy in individuals diagnosed with major depressive disorder: a non-randomized controlled trial. Front Psychiatry. 2023 Apr 28;14:1113956. doi: 10.3389/fpsyt.2023.1113956. eCollection 2023. PMID 37187863
- [Derived] Alavi N, Stephenson C, Yang M, Kumar A, Shao Y, Miller S, Yee CS, Stefatos A, Gholamzadehmir M, Abbaspour Z, Jagayat J, Shirazi A, Omrani M, Patel A, Patel C, Groll D. Feasibility and Efficacy of Delivering Cognitive Behavioral Therapy Through an Online Psychotherapy Tool for Depression: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Jun 16;10(6):e27489. doi: 10.2196/27489. PMID 33990076
- See also: Publication — https://www.frontiersin.org/journals/psychiatry/articles/10.3389/fpsyt.2023.1113956/full